CLINICAL TRIAL: NCT00123968
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA016-00-VP, Boosted by a Multiclade HIV-1 Recombinant Adenovirus-5 Vector Vaccine, VRC-HIVADV014-00-VP, in HIV Uninfected Adult Volunteers in East Africa
Brief Title: Safety of and Immune Response to an HIV-1 Vaccine (VRC-HIVDNA016-00-VP) and a Vaccine Booster (VRC-HIVADV014-00-VP) in HIV Uninfected East African Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 172; 10381 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2014-07

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (6):
- 1A (Experimental): Participants will receive a low dose of the adenovirus-vectored HIV vaccine or placebo at study entry
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-DILUENT013-DIL-VP
- 1B (Experimental): Participants will receive a higher dose of the adenovirus-vectored HIV vaccine or placebo at study entry
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-DILUENT013-DIL-VP
- 1C (Experimental): Participants will receive the DNA plasmid vaccine or placebo at study entry and Days 28 and 56. They will also receive either a low dose of the adenovirus-vectored HIV vaccine or placebo at Day 168.
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP; Biological: VRC-DILUENT013-DIL-VP; Biological: VRC-HIVADV014-00-VP placebo
- 1D (Experimental): Participants will receive the DNA plasmid vaccine or placebo at study entry and Days 28 and 56. They will also receive either a higher dose of the adenovirus-vectored HIV vaccine or placebo at Day 168.
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP; Biological: VRC-DILUENT013-DIL-VP; Biological: VRC-HIVADV014-00-VP placebo
- 2A (Experimental): Participants will receive the DNA plasmid vaccine at study entry and Days 28 and 56. They will also receive a low dose of the adenovirus-vectored HIV vaccine at Day 168.
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP; Biological: VRC-DILUENT013-DIL-VP
- 2B (Experimental): Participants will receive the DNA plasmid vaccine placebo at study entry and Days 28 and 56. They will also receive a the adenovirus-vectored HIV vaccine placebo at Day 168.
  Interventions: Biological: VRC-DILUENT013-DIL-VP; Biological: VRC-HIVADV014-00-VP placebo

INTERVENTIONS:
Biological: VRC-HIVDNA016-00-VP — 1x10^11 per unit vaccine administered intramuscularly via Bioinjector
  Arms: 1A; 1B; 1C; 1D; 2A
Biological: VRC-HIVADV014-00-VP — 4 mg administered intramuscularly via injection
  Arms: 1C; 1D; 2A
Biological: VRC-DILUENT013-DIL-VP — Administered intramuscularly via Bioinjector
  Other Names: VRC-HIVDNA016-00-VP placebo
Biological: VRC-HIVADV014-00-VP placebo — 4 mg administered intramuscularly via injection
  Arms: 1C; 1D; 2B

SUMMARY:
The purpose of the study is to determine the safety of and immune response to an investigational HIV vaccine, VRC-HIVDNA016-00-VP, and a vaccine booster, VRC-HIVADV014-00-VP, in HIV uninfected adults from Kenya, Tanzania, and Uganda.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development of a safe and effective vaccine that will prevent HIV infection. This study will evaluate the safety and immunogenicity of an experimental adenovirus-vectored multiclade HIV vaccine, VRC-HIVADV014-00-VP, followed with or without a similarly structured DNA plasmid HIV vaccine, VRC-HIVDNA016-00-VP. The DNA in both vaccines codes for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections in the world. HIV uninfected volunteers will be recruited in the East African nations of Kenya, Tanzania, and Uganda.

This study will comprise two parts, 1 and 2. Part 1 will enroll 144 participants who will be randomly assigned to one of four different groups:

* Group 1A participants will receive a low dose of the adenovirus-vectored HIV vaccine or placebo at study entry.
* Group 1B participants will receive a higher dose of the adenovirus-vectored HIV vaccine or placebo at study entry.
* Group 1C will receive the DNA plasmid vaccine or placebo at study entry and Days 28 and 56. They will also receive either a low dose of the adenovirus-vectored HIV vaccine or placebo at Day 168.
* Group 1D will receive the DNA plasmid vaccine or placebo at study entry and Days 28 and 56. They will also receive either a higher dose of the adenovirus-vectored HIV vaccine or placebo at Day 168.

Enrollment into Part 2 (Groups 2A and 2B) will begin after the completion of the safety data evaluation of Groups 3 and 4 and after Part A has been fully enrolled. Group 2A participants will receive the DNA plasmid vaccine or placebo at study entry and Days 28 and 56. They will also receive either a low dose of the adenovirus-vectored HIV vaccine or placebo at Day 168.

There will be 11 study visits over 14 to 16 months for Parts 1 and 2. All study visits will include a physical exam, medical and medication history, vital signs measurement, lymph node assessment, HIV and pregnancy counseling, and blood and urine collection. A home visit will also occur at study entry. A 3-day diary card to report side effects will be completed by participants at study entry and on Days 28, 56, 168, and 210.

There will be 14 study visits for Groups 3, 4, and 5; these visits will include the same tests and assessments as for Groups 1 and 2.

As per an amendment (dated December 19, 2005), follow-up for this study will be extended. The purpose for this extension is to examine in greater depth the efficacy of the vaccine. Specifically, investigators will be exploring whether there is a persistent immune response in participants who received the vaccine as well as if new or boosted responses to the adenovirus vaccine are persistent. The extended follow-up will last for 2 years with clinic visits every 4 months. During visits blood will be drawn for laboratory tests, including HIV testing. Participants will also be informed of ways to reduce their risk of contracting HIV. Two weeks after each visit, participants will be asked to come to the study site for a short post HIV test counseling visit. There will be a total of 6 visits per year, 3 follow-up visits, and 3 post HIV test counseling visits. There will be no more vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Willing to follow all the requirements of the study and available for follow-up for the duration of the study (14 to 16 months)
* Able and willing to provide informed consent
* Willing to undergo HIV testing and counseling and willing to receive HIV test results
* Willing to not engage in high-risk behavior for HIV infection during the study
* Willing to provide location and be visited at home
* Willing to be identified with picture identification for study purposes
* Willing to use acceptable forms of contraception
* Pregnant women and those with conditions which render phlebotomy volumes hazardous will be allowed to participate using a minimized phlebotomy schedule

Exclusion Criteria:

* HIV or HBV infection
* HIV vaccines in prior HIV vaccine trial
* Immunosuppressive or cytotoxic medications within the 6 months prior to study entry. Participants who have used corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for acute uncomplicated dermatitis are not excluded.
* Blood products within 120 days prior to study entry
* Immunoglobulin within 60 days prior to study entry
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Medically indicated subunit or killed vaccines or allergy treatment with antigen injections within 14 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Participated in high-risk behavior for HIV infection within 6 months prior to study entry. More information on this criterion can be found in the protocol.
* Serious adverse reactions to vaccines, such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Unstable asthma or asthma requiring emergent or urgent care, hospitalization, intubation, or oral or intravenous corticosteroids during the 2 years prior to study entry
* Diabetes mellitus type 1 or 2. Patients with gestational diabetes are not excluded.
* Thyroid disease, including removal of thyroid or disease requiring medication within 3 years prior to study entry
* Serious angioedema within 3 years prior to study entry or disease requiring medication within 2 years prior to study entry
* Uncontrolled hypertension
* Bleeding disorder
* Active syphilis
* Active cancer OR treated cancer that may recur during the duration of the study
* Seizure disorder. Participants who have had fever-related seizures prior to age 2 are not excluded.
* Absence of spleen OR partial or complete lack of splenic function
* Psychiatric condition that may interfere with the study, including past or present psychoses, bipolar disorder, or suicidal attempts
* Any medical, psychiatric, or social condition that, in the opinion of the investigator, may interfere with the study
* Any occupational or other responsibility that, in the opinion of the investigator, may interfere with the study
* Pregnancy, breastfeeding, or plan to become pregnant
* Any occupational or other responsibility that, in the opinion of the investigator, may interfere with the study
* Incapacitating illness precluding clinic visits
* Unable to provide informed consent
* Prisoners will not be enrolled while incarcerated and if enrolled prior to incarceration, will not be followed while in confinement. Re-consent will not be required upon release from prison.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2006-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms | Throughout study
Systemic reactogenicity signs and symptoms | Throughout study
Laboratory measures of safety | Throughout study
Adverse and serious adverse experiences | Throughout study
Unfractionated IFN-gamma ELISPOT responses to HIV-1 | At Day 196
CD4+ and CD8+ T cell responses to HIV-1, as measured by flow cytometry-based intracellular cytokine staining (ICS) assay | At Day 196

CONTACTS AND LOCATIONS:
Overall Officials: Merlin Robb, MD, Study Chair — US Military HIV Research Program
Locations (3):
- Kenya Med. Research Inst./Walter Reed Project, Clinical Research Centre, Off Hospital Road. Kericho, Kericho, Kenya
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) CRS, Mbeya, Tanzania
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

REFERENCES:
- [Background] Esparza J, Osmanov S. HIV vaccines: a global perspective. Curr Mol Med. 2003 May;3(3):183-93. doi: 10.2174/1566524033479825. PMID 12699356
- [Background] Gaschen B, Taylor J, Yusim K, Foley B, Gao F, Lang D, Novitsky V, Haynes B, Hahn BH, Bhattacharya T, Korber B. Diversity considerations in HIV-1 vaccine selection. Science. 2002 Jun 28;296(5577):2354-60. doi: 10.1126/science.1070441. PMID 12089434
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Derived] Kibuuka H, Kimutai R, Maboko L, Sawe F, Schunk MS, Kroidl A, Shaffer D, Eller LA, Kibaya R, Eller MA, Schindler KB, Schuetz A, Millard M, Kroll J, Dally L, Hoelscher M, Bailer R, Cox JH, Marovich M, Birx DL, Graham BS, Michael NL, de Souza MS, Robb ML. A phase 1/2 study of a multiclade HIV-1 DNA plasmid prime and recombinant adenovirus serotype 5 boost vaccine in HIV-Uninfected East Africans (RV 172). J Infect Dis. 2010 Feb 15;201(4):600-7. doi: 10.1086/650299. PMID 20078213
- [Derived] Kibuuka H, Guwatudde D, Kimutai R, Maganga L, Maboko L, Watyema C, Sawe F, Shaffer D, Matsiko D, Millard M, Michael N, Wabwire-Mangen F, Robb M. Contraceptive use in women enrolled into preventive HIV vaccine trials: experience from a phase I/II trial in East Africa. PLoS One. 2009;4(4):e5164. doi: 10.1371/journal.pone.0005164. Epub 2009 Apr 10. PMID 19360102